CLINICAL TRIAL: NCT06763900
Title: Comparison of the Effectiveness of Corticotomy-Assisted Different Miniplate and Intermaxillary Elastic Applications After Growth Spurt in Individuals with Skeletal Class III Malocclusion
Brief Title: Corticotomy-Assisted Class III Elastic Applications
Acronym: CACIIIEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ahmet Yağcı, Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDH-2022-11536
Record Dates: First submitted 2023-06-07; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2023-06

CONDITIONS: Class III Malocclusion
Keywords: Class III Malocclusion; Miniplates; Corticotomy; Skeletal Anchorage; Class III Elastics
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: Twenty patients aged between 13-15 years were randomly divided into three groups. In acrylic splint group (AS) and palatal miniscrew group (MS), an acrylic splint containing hooks in the upper molar region was prepared and cemented. In the MS group, two miniscrews were used in the palatal region for additional anchorage. An incomplete Le Fort 1 osteotomy was performed in all patients to free the maxilla. Miniplates were placed vertically between the mandibular canine and first premolar in all groups, and horizontally under the osteotomy line in the maxillary molar region in miniplate group (MP). Class III elastics were applied 5 days after the surgery. Treatment was continued until a positive overjet was achieved. Cephalometric radiographs were taken at the beginning of treatment (T0) and at the end of the protraction period (T1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Miniplate Group (MP) (Experimental): An incomplete Le Fort 1 osteotomy was performed in all patients to free the maxilla. Miniplates were placed vertically between the mandibular canine and first premolar in all groups, and horizontally under the osteotomy line in the maxillary molar region. Class III elastics were applied 5 days after the surgery. Treatment was continued until a positive overjet was achieved. Cephalometric radiographs were taken at the beginning of treatment (T0) and at the end of the protraction period (T1).
  Interventions: Device: Skeletal anchorage and intermaxillary elastic assisted maxillary protraction
- Acrylic Splint Group (AS) (Experimental): An acrylic splint containing hooks in the upper molar region was prepared and cemented to the upper dentition. An incomplete Le Fort 1 osteotomy was performed in all patients to free the maxilla. Miniplates were placed vertically between the mandibular canine and first premolar in all groups, and horizontally under the osteotomy line in the maxillary molar region in miniplate group (MP). Class III elastics were applied 5 days after the surgery. Treatment was continued until a positive overjet was achieved. Cephalometric radiographs were taken at the beginning of treatment (T0) and at the end of the protraction period (T1).
  Interventions: Device: Skeletal anchorage and intermaxillary elastic assisted maxillary protraction
- Palatal Miniscrew Supported Acrylic Splint Group (MS) (Experimental): An acrylic splint containing hooks in the upper molar region was prepared and cemented to the upper dentition. Two miniscrews were used in the palatal region for additional anchorage. An incomplete Le Fort 1 osteotomy was performed in all patients to free the maxilla. Miniplates were placed vertically between the mandibular canine and first premolar in all groups, and horizontally under the osteotomy line in the maxillary molar region in miniplate group (MP). Class III elastics were applied 5 days after the surgery. Treatment was continued until a positive overjet was achieved. Cephalometric radiographs were taken at the beginning of treatment (T0) and at the end of the protraction period (T1).
  Interventions: Device: Skeletal anchorage and intermaxillary elastic assisted maxillary protraction

INTERVENTIONS:
Device: Skeletal anchorage and intermaxillary elastic assisted maxillary protraction — maxillary protraction with corticotomy-assisted different miniplate and intermaxillary elastic applications after growth spurt in patients with skeletal Class III malocclusion

SUMMARY:
This prospective randomized clinical study aimed to evaluate the effectiveness of corticotomy-assisted maxillary protraction with three different miniplate and intermaxillary elastic applications after corticotomy in patients with skeletal Class III malocclusion.

DETAILED DESCRIPTION:
In acrylic splint group (AS) and palatal miniscrew group (MS), an acrylic splint containing hooks in the upper molar region was prepared and cemented. In the MS group, two miniscrews were used in the palatal region for additional anchorage. An incomplete Le Fort 1 osteotomy was performed in all patients to free the maxilla. Miniplates were placed vertically between the mandibular canine and first premolar in all groups, and horizontally under the osteotomy line in the maxillary molar region in miniplate group (MP). Class III elastics were applied 5 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Class III malocclusion
* ANB angle between 0 and -4°
* normal or horizontal growth pattern
* anterior crossbite or edge-to-edge incisor relationship
* permanent dentition

Exclusion Criteria:

* requirement for maxillary expansion
* pseudo-Class III malocclusion
* inadequate oral hygiene
* missing tooth in the upper dentition

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Maxillomandibular sagittal changes | Through study completion, an avarage of 6 months
  Investigation of Angular changes in SNA (°), SNB (°), ANB (°) measurements. Investigation of Distance changes in Wits (mm), A-Na Perp (mm), Co-A (mm), A-VRL (mm), and B-VRL (mm) measurements.
Vertical changes | Through study completion, an avarage of 6 months
  Investigation of Angular changes in Y-axis angle (°), SN-GoGN (°), SN-PP (°), Jarabak ratio measurements.
  Investigation of Distance changes in A-HRL (mm) measurement.
Dentoalveolar changes | Through study completion, an avarage of 6 months
  Investigation of Angular changes in U1-SN (°), U1-PP (°), IMPA (°) measurements.
  Investigation of Distance changes in Overjet (mm), Overbite (mm), U1-VRL (mm), and U6-VRL (mm) measurements.
Soft tissue changes | Through study completion, an avarage of 6 months
  Investigation of Angular changes in soft tissue convexity (°), NA-Pog (°) measurements.
  Investigation of Distance changes in VRL-prn (mm), VRL-Is (mm), VRL-li (mm), VRL-pog (mm), and ANS-Me (mm) measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YAĞCI, Professor, Study Director
Locations (1):
- Erciyes University Faculty of Dentistry, Department of Orthodontics, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Clerck HJ, Cornelis MA, Cevidanes LH, Heymann GC, Tulloch CJ. Orthopedic traction of the maxilla with miniplates: a new perspective for treatment of midface deficiency. J Oral Maxillofac Surg. 2009 Oct;67(10):2123-9. doi: 10.1016/j.joms.2009.03.007. No abstract available. PMID 19761906
- [Background] Yilmaz HN, Garip H, Satilmis T, Kucukkeles N. Corticotomy-assisted maxillary protraction with skeletal anchorage and Class III elastics. Angle Orthod. 2015 Jan;85(1):48-57. doi: 10.2319/121513-921.1. PMID 24913740
- [Background] Willmann JH, Nienkemper M, Tarraf NE, Wilmes B, Drescher D. Early Class III treatment with Hybrid-Hyrax - Facemask in comparison to Hybrid-Hyrax-Mentoplate - skeletal and dental outcomes. Prog Orthod. 2018 Oct 22;19(1):42. doi: 10.1186/s40510-018-0239-8. PMID 30345472
- [Background] Kircelli BH, Pektas ZO. Midfacial protraction with skeletally anchored face mask therapy: a novel approach and preliminary results. Am J Orthod Dentofacial Orthop. 2008 Mar;133(3):440-9. doi: 10.1016/j.ajodo.2007.06.011. PMID 18331946
- [Background] Sar C, Sahinoglu Z, Ozcirpici AA, Uckan S. Dentofacial effects of skeletal anchored treatment modalities for the correction of maxillary retrognathia. Am J Orthod Dentofacial Orthop. 2014 Jan;145(1):41-54. doi: 10.1016/j.ajodo.2013.09.009. PMID 24373654